CLINICAL TRIAL: NCT07235683
Title: Combination Letermovir and Standard of Care Antiviral for Enhanced Antiviral Response in Cytomegalovirus Infection in Lung Transplant Recipients: A Pilot Trial
Brief Title: Combination Letermovir and Standard of Care Antiviral for Enhanced Antiviral Response in Cytomegalovirus Infection in Lung Transplant Recipients
Acronym: CLEAR-CMV
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-5760
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: CMV; Lung Transplant Recipient
Keywords: CMV Disease; Lung Transplant
MeSH Terms: interventions — letermovir; Valganciclovir; Ganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOC antiviral plus placebo (Placebo Comparator): Patients will receive the standard of care (SOC) antiviral therapy along with a placebo drug. The placebo drug will be administered for three weeks, while the SOC antiviral duration and dosage will be at the discretion of the treating physician.
  Interventions: Drug: Placebo; Drug: Valganciclovir/Ganciclovir
- SOC antiviral plus letermovir active drug (Experimental): Patients will receive the standard of care (SOC) antiviral therapy in combination with letermovir. The letermovir active drug will be administered for three weeks, while the SOC antiviral treatment duration and dosage will be at the discretion of the treating physician.
  Interventions: Drug: Letermovir; Drug: Valganciclovir/Ganciclovir

INTERVENTIONS:
Drug: Letermovir — Letermovir (480mg) will be given orally as a loading dose every 12 hours for the first 24 hours, then one tablet per day for a total treatment duration of 21 days. Letermovir treatment will be started within 72 hours of starting SOC antiviral treatment as per the decision of the treating physician.
  Arms: SOC antiviral plus letermovir active drug
Drug: Placebo — Placebo will be dosed the same as letermovir: one tablet every 12 hours for the first 24 hours, then one tablet per day for total treatment duration of 21 days.
  Arms: SOC antiviral plus placebo
Drug: Valganciclovir/Ganciclovir — Ganciclovir or its oral prodrug, valganciclovir will be administered as the standard of care antiviral therapy. Its duration will be at the discretion of the treatment physician but is typically given until clearance of viremia. The clinical definition of viral clearance is one negative viral load or two viral loads one week apart that are <200 IU/mL

SUMMARY:
The primary objective of the CLEAR-CMV trial is to evaluate the efficacy of letermovir therapy plus standard of care (SOC) antiviral compared to SOC plus placebo in achieving clearance of CMV viremia by week 3 in lung transplant recipients with active CMV infection.

DETAILED DESCRIPTION:
Lung transplant recipients are particularly susceptible to CMV infection due to intensive immunosuppressive regimens required to prevent graft rejection. CMV viremia is associated with increased morbidity, including CMV pneumonitis, and may contribute to chronic lung allograft dysfunction (CLAD).Approximately 30-50% of lung transplant recipients develop CMV infection within the first year post-transplant, with higher rates in CMV-seronegative recipients receiving organs from seropositive donors (D+/R-).

Current standard treatment for CMV infection in transplant recipients involves ganciclovir or its oral prodrug, valganciclovir, which inhibit CMV DNA polymerase. While effective, prolonged use is associated with toxicities, including myelosuppression, and the emergence of resistant strains in some cases. Letermovir, a novel antiviral targeting the CMV terminase complex, has shown efficacy in CMV prophylaxis in hematopoietic stem cell transplant recipients, and in kidney transplant recipients. It has now been extensively studied for use in prophylaxis but there are limited data in treatment. It is an attractive drug in transplant recipients because it has an excellent safety profile and requires no dose adjustment for renal dysfunction. However, data on the use of letermovir for treatment (as opposed to prophylaxis) are more limited. A multicenter study of letermovir use for treatment showed reasonable response rates especially in patients with low viral loads. The use of combination therapy for CMV treatment represents an attractive option, as there is extensive experience with other viruses (e.g. HIV , HCV) to show that this strategy leads to improved response rates and lessens the emergence of antiviral resistance. The use of ganciclovir plus letermovir is attractive because they target two different viral enzymes and both have oral options facilitating outpatient treatment. The most recently published international CMV consensus guidelines reports that the use of combination antiviral therapy is a key research need.

The investigators plan to conduct a pilot trial to determine the efficacy of letermovir plus standard of care (SOC) antiviral therapy in clearing CMV infection. The trial will be conducted in compliance with the protocol, Good Clinical Practices (GCP) and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a lung transplant.
* Has confirmed CMV viremia with a viral load ≥ 1000 IU/mL and will receive or has just started SOC antiviral treatment in the past 72h as per the decision of the treating physician.

Exclusion Criteria:

* Renal failure with Creatinine clearance <15 mL/min or requiring dialysis
* Severe hepatic impairment (Child-Pugh Class C)
* Participating in another interventional clinical trial
* Combined transplant (e.g heart-lung, lung-liver)
* Known allergy or contraindication to any of the antiviral medications
* Known antiviral resistance.
* Patient receiving cyclosporin, pimozide or ergot alkaloids (due to significant drug interaction with letermovir).
* Patient receiving or expected to receive CMV immunoglobulin or IVIG during the initial three week treatment phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving clearance of CMV viremia by week 3, as measured by quantitative PCR. | From time of enrollment until 3 weeks after enrolment
  Viral clearance is described by a plasma CMV viral load < 200 IU/mL, the UHN clinically used threshold

SECONDARY OUTCOMES:
Proportion of patients achieving an undetectable viral load | At week 3 and by month 6 after enrolment
  The limit of detection for plasma CMV viral load is 35 IU/mL
Proportion of patients achieving CMV viral load <137 IU/mL (lower limit of quantification of the assay) | At week 3 from enrolment and at 6 months
  Lower limit of viral quantitation
Time to clearance of CMV viremia | From enrolment until clearance of CMV viremia, up to 6 months after enrolment
  Clearance of CMV viremia is defined as plasma CMV viral load < 200 IU/mL as measured by quantitative PCR
Time to resolution of symptoms if present | From enrolment until clearance of symptoms, up to 6 months after enrolment
Development of antiviral resistance | From enrolment until up to 6 months after enrolment
  Incidence of antiviral resistance development to letermovir or SOC antivirals at the discretion of the treatment physician
Incidence of adverse events | From enrolment until up to 6 months after enrolment
  Incidence of adverse effects (e.g., myelosuppression, renal dysfunction) will be recorded for the duration of the study.
Proportion of patients with clinically significant CMV recurrence within 6months, as determined by quantitative PCR or symptomatic CMV disease | From enrollment until 6 months.
  Clinically significant CMV recurrence will be determined by a qPCR viral load ≥1000 IU/mL or symptomatic CMV disease
Monthly enrollment rate as a measure of recruitment feasibility | From start of enrollment until up to 6 months after the final patient is enrolled
  The investigators will aim for a target enrollment rate of 2 participants per month

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada